CLINICAL TRIAL: NCT03162107
Title: Promoting Engagement in the Drug Resistant TB/HIV Care Continuum in South Africa PRAXIS Study (PRospective Study of Adherence in M/XDR-TB Implementation Science)
Brief Title: Promoting Engagement in the Drug Resistant TB/HIV Care Continuum in South Africa
Acronym: PRAXIS
Status: Completed | Type: Observational
Sponsor: Centre for the AIDS Programme of Research in South Africa (Network)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Dr Nesri Padayatchi, Deputy Director, Centre for the AIDS Programme of Research in South Africa
Other Study IDs: CAP 086
Record Dates: First submitted 2017-03-24; First posted 2017-05-22 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Patient Non-compliance
Keywords: adherence; HIV; MDR/XDR TB; Health Care Worker
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Hair samples PBMCs TB Isolates
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goals of this research are to understand adherence and retention in care for multi-and extensively drug-resistant tuberculosis (M/XDR-TB) patients using a mixed methods approach.

DETAILED DESCRIPTION:
Tuberculosis (TB) remains the leading cause of morbidity and mortality worldwide among people living with HIV. Globally, incidence of multidrug-resistant tuberculosis (MDR-TB) and extensively drug resistant tuberculosis (XDR-TB), the most drug-resistant forms of TB, has approximately doubled over the past fifteen years. Nowhere has this increased incidence generated more concern than in South Africa where interactions between TB and generalized HIV epidemics are causing 'explosive' TB incidence and case-fatality threatening to undermine the progress reached with antiretroviral therapy (ART).

Medication adherence, a key predictor of outcomes in multi-and extensively drug-resistant tuberculosis (M/XDR-TB) and HIV treatment, is understudied in high burden TB/HIV settings. Patient losses during transitions in the care continuum are frequent, increase mortality and limit control of the linked epidemics. Demands of M/XDR-TB HIV treatment are severe including extraordinary pill burden, severe adverse effects, lengthy treatment, isolation and stigma with few parallels in modern medicine.

This is a prospective observational cohort study for patients newly diagnosed with M/XDR-TB initiating treatment. A mixed method approach will be employed to address the complex research questions of distilling determinants of barriers and facilitators to both TB medications and ART; this study will employ complementary qualitative and quantitative methodologies for assessing differential adherence to TB medications and ART.

A sub-set of patients and health care workers will be approached for participation in focus group discussions.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Mycobacterium Tuberculosis (MTB) culture positive with at least isoniazid and rifampicin resistance OR

   Molecular drug susceptibility test confirming resistance to at least isoniazid and rifampicin OR

   Polymerase chain reaction test (GeneXpert MTB/RIF) result showing MTB positive and RIF resistance. Patients enrolled with only a GeneXpert MTB/RIF result will be withdrawn if their subsequent susceptibility test or molecular drug susceptibility test reveals rifampicin monoresistance.
3. Initiating treatment for M/XDR-TB which includes at least 2 new medications
4. Have capacity for informed consent
5. HIV Positive Patients: on antiretroviral therapy (ART) or initiating ART within the following 4 weeks as per clinician recommendation

Exclusion Criteria:

1. Pregnancy
2. Prisoners
3. Discretion of the Investigator of Record or clinician

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult patients with newly diagnosed active pulmonary multi- and extremely-drug resistance tuberculosis (M/XDR-TB) (≥ 18 years old), admitted for routine care at King DinuZulu Hospital in Durban, South Africa will be approached for enrollment. Only patients with capacity for consent will be included in the study. Healthcare workers will be approached for participation in focus group discussions.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
Medication adherence based on electronic monitoring | 6 months
  An electronic monitoring system (e.g., Wisepill technologies) will be used to measure adherence to antiretroviral therapy and treatment of multi- and extremely-drug resistant tuberculosis.

SECONDARY OUTCOMES:
Medication adherence based on self-report | 6 months
  Quantitative adherence will be measured using 30 day and 7 day recall. Average adherence to both antiretroviral therapy and tuberculosis treatment will be calculated for each patient
Sociomedical risk factors associated with six-month adherence to ART or TB medications | 6 months
  Barriers and facilitators to medication adherence and retention in care for M/XDR-TB HIV patients will be identified through in-depth interviews and focus group discussions with patients and health care workers. To identify sociomedical risk factors associated with six-month adherence to ART or TB medications we will first identified risk factors associated with adherence in bivariate analysis and then multiple logistic regression models will be constructed including variables which are statistically significant and/or associated with >10% change in effect measure.

CONTACTS AND LOCATIONS:
Overall Officials: Nesri Padayatchi, MBChB, Principal Investigator — Centre for the AIDS Programme of Research in South Africa
Locations (1):
- King Dinuzulu Hospital, Durban, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bateman M, Wolf A, Chimukangara B, Brust JCM, Lessells R, Amico R, Boodhram R, Singh N, Orrell C, Friedland G, Naidoo K, Padayatchi N, O'Donnell MR. Adherence Measured Using Electronic Dose Monitoring is Associated with Emergent Antiretroviral Resistance and Poor Outcomes in People with Human Immunodeficiency Virus/AIDS and Multidrug-Resistant Tuberculosis. Clin Infect Dis. 2022 Oct 29;75(9):1489-1496. doi: 10.1093/cid/ciac232. PMID 35352097